CLINICAL TRIAL: NCT02273206
Title: Collaborative Care to Reduce Depression and Increase Cancer Screening Among Low-Income Urban Women Project
Brief Title: Collaborative Care to Reduce Depression and Increase Cancer Screening Among Low-Income Urban Women
Acronym: PCM3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Directors Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IH-12-11-4522
Record Dates: First submitted 2014-10-17; First posted 2014-10-23 (Estimated); Results first posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-02

CONDITIONS: Depression; Breast Cancer Screening; Cervical Cancer Screening; Colorectal Cancer Screening
Keywords: Depression; Breast Cancer Screening; Cervical Cancer Screening; Colorectal Cancer Screening
MeSH Terms: conditions — Depression | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prevention Care Management for Cancer Screening (Active Comparator): The Care Manager will focus on cancer screening, providing education, patient navigation, and motivational support to overcome screening barriers and form favorable attitudes towards screening.
  Interventions: Behavioral: Prevention Care Management for Cancer Screening
- Prevention Care Management for Depression and Cancer Screening (Experimental): The Care Manager will provide depression care management and motivational support (supportive counseling) and act as a critical link between primary care, mental health care provider, and the patients, helping to develop and implement a treatment plan.
  In addition, the Care Manager will work with participants on cancer screening, providing education, patient navigation, and motivational support to overcome screening barriers and form favorable attitudes towards screening.
  Interventions: Behavioral: Prevention Care Management for Depression and Cancer Screening; Behavioral: Prevention Care Management for Cancer Screening

INTERVENTIONS:
Behavioral: Prevention Care Management for Depression and Cancer Screening
  Other Names: Collaborative Care Intervention (CCI)
  Arms: Prevention Care Management for Depression and Cancer Screening
Behavioral: Prevention Care Management for Cancer Screening
  Other Names: Prevention Care Manager (PCM)

SUMMARY:
Bronx County, New York is the poorest urban county in the U.S.A., and residents are almost entirely Latino or African American. Cancer is the leading cause of premature death in the Bronx, with morality rates significantly higher than for New York City as a whole. Low-income/minority populations are more likely to be diagnosed with preventable and late-stage cancers than the general population, in part, due to lower screening rates. While research has addressed screening barriers in low-income/minority groups, depression, a common,potentially critical barrier, has received scant attention. Research suggests that depressed women are less likely to engage in cancer screening, especially mammography and Pap testing. The link between mental health and cancer screening is particularly important to address in the Bronx, which has the highest rates of self-reported serious psychological distress (a measure closely related to depression) in New York City. Depression affects almost 1 in 4 minority women, and while minorities often seek help for depression in primary care, primary care depression management often does not meet evidence-based standards. Drawing on the expertise and close collaboration of Bronx medical and social service providers and patient stakeholders, this study will determine whether a collaborative care intervention that addresses both depression and cancer screening needs simultaneously among women ages 50-64 is more effective at improving cancer screening and patient-reported outcomes for women with depression than an existing evidence-based cancer screening intervention alone.

To achieve this, the investigators will compare the effectiveness of these two interventions using a randomized controlled trial (RCT). In partnership with six Bronx Federally Qualified Health Centers (FQHCs), the investigators will recruit approximately 800 women ages 50-64 who screen positive for depression and are non-adherent with recommended cervical, breast, and/or colorectal cancer screenings. The investigators specific aims are to: 1) compare the impact of the two interventions on patient-reported outcomes, including cancer screening knowledge and attitudes, self-efficacy, depression-related stigma, provider referrals, participation in mental health care, medication adherence, quality of life, satisfaction with care and treatment decisions, and depression; 2) compare the effectiveness of the two interventions in increasing breast, cervical, and colorectal cancer screening; 3) determine whether reducing depression increases the likelihood that low-income women 50-64 will receive cancer screening; 4) determine whether effectiveness of the two interventions in increasing cancer screening varies according to patient characteristics, such as duration of depression, presence of other chronic conditions, and obesity.

This study is designed to increase the investigators understanding of how to enhance primary care systems' ability to improve a range of outcomes related to cancer screening and depression among low-income minority women, and how to best support this population in making cancer-screening decisions.

ELIGIBILITY:
Inclusion Criteria:

* Resident of the Bronx
* Overdue for breast, cervical or colorectal cancer screening
* Screen positive for depression
* No cancer diagnosis within the past six months

Ages: 50 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 802 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Weiss, PhD, Principal Investigator — The Leukemia and Lymphoma Society; Jonathan N Tobin, PhD, Principal Investigator — Clinical Directors Nework; Andrea Cassells, MPH, Study Director — Clinical Directors Network
Locations (8):
- United States (8):
  - Lincoln Ambulatory Care Practice, The Bronx, New York
  - Morrissania Diagnostic and Treatment Center, The Bronx, New York
  - Morris Heights Health Center, The Bronx, New York
  - Segundo Ruiz Belvis Diagnostic and Treatment Center, The Bronx, New York
  - BronwWorks, The Bronx, New York
  - Urban Health Plan, The Bronx, New York
  - Montefiore Family Care Center, The Bronx, New York
  - Good Shepherd Service, The Bronx, New York

REFERENCES:
- [Derived] Tobin JN, Cassells A, Weiss E, Lin TJ, Holder T, Carrozzi G, Barsanti F, Morales A, Maling A, Espejo M, Ascher A, Gilbert E, Casiano L, O-Hara-Cicero E, Weed J, Dietrich A. Integrating Cancer Screening and Mental Health Services in Primary Care: Protocol and Baseline Results of a Patient-Centered Outcomes Intervention Study. J Health Care Poor Underserved. 2021;32(4):1907-1934. doi: 10.1353/hpu.2021.0173. PMID 34803050

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Among the 802 participants who were recruited for the study, 759 completed the baseline assessment and were randomized to one of the two intervention groups. Two participants were found to be ineligible after randomization and were excluded; as a result, 757 participants are included in the analyses.
Groups:
- Collaborative Care Intervention (CCI): Participants assigned to the CCI group received the Prevention Care Management (PCM) intervention, as well as motivational support to initiate or follow up on mental health treatment and linkages to social support services.
- Prevention Care Management (PCM) Intervention: The PCM intervention consisted of cancer screening telephone support, including education, patient navigation, and motivational interviewing to overcome barriers to screening.
Period: Overall Study
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM) Intervention
Started | 378 | 379
Completed | 353 | 337
Not Completed | 25 | 42

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM) Intervention | Total
Number analyzed (Participants) | 378 | 379 | 757
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (4.3) | 55.8 (4.2) | 56.0 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 378 | 379 | 757
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 289 | 301 | 590
  Not Hispanic or Latino | 89 | 78 | 167
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Some participants did not provide a response for this question.
  Participants
    number analyzed (Participants) | 376 | 379 | 755
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 82 | 67 | 149
    White | 19 | 12 | 31
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 275 | 300 | 575
Region of Enrollment [Number; unit: participants]
  United States | 378 | 379 | 757
Primary Language [Count of Participants; unit: Participants]
  English | 163 | 167 | 330
  Spanish | 215 | 212 | 427
Country of Birth [Count of Participants; unit: Participants] — Population: Some participants did not provide a response for this question.
  Participants
    Born in U.S.: number analyzed (Participants) | 377 | 377 | 754
    Born in U.S. | 142 | 154 | 296
    Born outside of U.S.: number analyzed (Participants) | 377 | 377 | 754
    Born outside of U.S. | 235 | 223 | 458
Marital Status [Count of Participants; unit: Participants] — Population: Some participants did not provide a response for this question.
  Participants
    Married/cohabitating: number analyzed (Participants) | 376 | 378 | 754
    Married/cohabitating | 95 | 95 | 190
    Single/divorced/widowed/separated: number analyzed (Participants) | 376 | 378 | 754
    Single/divorced/widowed/separated | 271 | 274 | 545
    Other: number analyzed (Participants) | 376 | 378 | 754
    Other | 10 | 9 | 19
Education [Count of Participants; unit: Participants] — Population: Some participants did not provide a response for this question.
  Participants
    Less than 8 years: number analyzed (Participants) | 376 | 376 | 752
    Less than 8 years | 89 | 81 | 170
    8-11 years: number analyzed (Participants) | 376 | 376 | 752
    8-11 years | 113 | 131 | 244
    Completed High School: number analyzed (Participants) | 376 | 376 | 752
    Completed High School | 90 | 82 | 172
    Post High School and higher: number analyzed (Participants) | 376 | 376 | 752
    Post High School and higher | 84 | 82 | 166
Employment [Count of Participants; unit: Participants]
  Employed | 76 | 78 | 154
  Unemployed | 102 | 108 | 210
  Homemaker | 61 | 59 | 120
  Other | 139 | 134 | 273
Household income [Count of Participants; unit: Participants] — Population: Some participants did not provide a response for this question.
  Participants
    $0 to $9,999: number analyzed (Participants) | 374 | 373 | 747
    $0 to $9,999 | 258 | 242 | 500
    $10,000 to $14,999: number analyzed (Participants) | 374 | 373 | 747
    $10,000 to $14,999 | 42 | 69 | 111
    $15,000 or more: number analyzed (Participants) | 374 | 373 | 747
    $15,000 or more | 74 | 62 | 136
Insurance [Count of Participants; unit: Participants] — Population: Some participants did not provide a response for this question.
  Participants
    Medicaid + Medicare: number analyzed (Participants) | 377 | 379 | 756
    Medicaid + Medicare | 32 | 32 | 64
    Medicaid: number analyzed (Participants) | 377 | 379 | 756
    Medicaid | 275 | 285 | 560
    Medicare: number analyzed (Participants) | 377 | 379 | 756
    Medicare | 17 | 12 | 29
    Employer: number analyzed (Participants) | 377 | 379 | 756
    Employer | 12 | 17 | 29
    No insurance: number analyzed (Participants) | 377 | 379 | 756
    No insurance | 41 | 33 | 74
Years receiving care at the community health center before consent [Count of Participants; unit: Participants] — Population: Some participants did not provide a response for this question.
  Participants
    < 3: number analyzed (Participants) | 377 | 377 | 754
    < 3 | 126 | 138 | 264
    ≥ 3: number analyzed (Participants) | 377 | 377 | 754
    ≥ 3 | 251 | 239 | 490
Patient Health Questionnaire-9 (PHQ9) Score Group [Count of Participants; unit: Participants] — Population: Some participants did not provide a response for this question.
  Participants
    Mild Depression (5-9): number analyzed (Participants) | 377 | 379 | 756
    Mild Depression (5-9) | 104 | 104 | 208
    Moderate Depression (10-14): number analyzed (Participants) | 377 | 379 | 756
    Moderate Depression (10-14) | 159 | 147 | 306
    Moderately Severe Depression (15-19): number analyzed (Participants) | 377 | 379 | 756
    Moderately Severe Depression (15-19) | 80 | 102 | 182
    Severe Depression (20-27): number analyzed (Participants) | 377 | 379 | 756
    Severe Depression (20-27) | 34 | 26 | 60
Cancer Screening [Count of Participants; unit: Participants]
  Up to date for Colorectal Cancer Screening | 83 | 102 | 185
  Up to date for Breast Cancer Screening | 166 | 159 | 325
  Up to date for Cervical Cancer Screening | 160 | 158 | 318
Cancer history [Count of Participants; unit: Participants] — Population: Some participants did not provide a response for this question.
  Participants
    number analyzed (Participants) | 377 | 376 | 753
    (all) | 28 | 32 | 60
Hysterectomy [Count of Participants; unit: Participants] — Population: Some participants did not provide a response for this question.
  Participants
    number analyzed (Participants) | 377 | 374 | 751
    (all) | 84 | 83 | 167
Smoking Status [Count of Participants; unit: Participants] — Population: Electronic health record data for this measure is not available for all participants.
  Participants
    Current: number analyzed (Participants) | 308 | 320 | 628
    Current | 92 | 89 | 181
    Former: number analyzed (Participants) | 308 | 320 | 628
    Former | 50 | 53 | 103
    Never: number analyzed (Participants) | 308 | 320 | 628
    Never | 166 | 178 | 344
Comorbid Condition- Asthma [Count of Participants; unit: Participants] — Population: Electronic health record data for this measure is not available for all participants.
  Participants
    number analyzed (Participants) | 377 | 378 | 755
    (all) | 124 | 123 | 247
Comorbid Condition- Hypertension [Count of Participants; unit: Participants] — Population: Electronic health record data for this measure is not available for all participants.
  Participants
    number analyzed (Participants) | 377 | 378 | 755
    (all) | 242 | 245 | 487
Comorbid Condition- Hyperlipidemia [Count of Participants; unit: Participants] — Population: Electronic health record data for this measure is not available for all participants.
  Participants
    number analyzed (Participants) | 377 | 378 | 755
    (all) | 220 | 209 | 429
Comorbid Condition- Diabetes [Count of Participants; unit: Participants] — Population: Electronic health record data for this measure is not available for all participants.
  Participants
    number analyzed (Participants) | 377 | 378 | 755
    (all) | 157 | 152 | 309

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Colorectal, Breast, and Cervical Cancer Screening Up to Date Status
Description: Comparison of the proportion of patients who were up to date for colorectal cancer, breast cancer and cervical cancer screenings before and after the intervention. (Chart Review)
Time Frame: Baseline - 12 months
Measure: Number; unit: Percentage (%) of Participants
Groups:
- Prevention Care Management (PCM): The PCM intervention consisted of cancer screening telephone support, including education, patient navigation, and motivational interviewing to overcome barriers to screening
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM)
Number analyzed (Participants) | 378 | 379
Percentage (%) of Participants
  Colorectal Cancer Screening - Baseline | 22.0 | 26.9
  Colorectal Cancer Screening - Follow Up | 56.9 | 52.8
  Breast Cancer Screening - Baseline | 43.9 | 42.0
  Breast Cancer Screening - Follow Up | 66.7 | 66.8
  Cervical Cancer Screening - Baseline | 42.3 | 41.7
  Cervical Cancer Screening - Follow Up | 61.6 | 64.6
Statistical Analysis 1: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Colorectal Cancer Screening Intervention Arm Difference; Test type: Superiority; p = 0.2562, Chi-squared; p<0.05
Statistical Analysis 2: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Breast Cancer Screening Intervention Arm Difference; Test type: Superiority; p = 0.9795, Chi-squared; p<0.05
Statistical Analysis 3: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Cervical Cancer Screening Intervention Arm Difference; Test type: Superiority; p = 0.3917, Chi-squared; p<0.05

2. Primary Outcome: Assessment of Colorectal Cancer Screening Up to Date Status After Intervention
Description: Multivariate logistic regression model was used to assess which factors contributed to colorectal cancer screening up to date status.
Time Frame: Baseline - 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM)
Number analyzed (Participants) | 378 | 379
percentage of participants
  Up to Date at Baseline | 22.0 | 26.9
  Up to Date at Follow Up | 56.9 | 52.8
Statistical Analysis 1: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Test type: Superiority — Test the coefficient for intervention; p = 0.0677, Regression, Logistic — Treatment Group (CCI vs PCM); p<0.05; Odds Ratio (OR) = 1.346, 95% CI 2-sided [0.979 to 1.851] — In the logistic regression model, adjustments were made for PHQ9 at baseline, improvement of depression by one level, baseline colorectal cancer up to date status, age, and income

3. Primary Outcome: Assessment of Breast Cancer Screening Up to Date Status After Intervention
Description: Multivariate logistic regression model was used to assess which factors contributed to breast cancer screening up to date status
Time Frame: Baseline - 12 months
Measure: Number; unit: Percentage of Participants
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM)
Number analyzed (Participants) | 378 | 379
Percentage of Participants
  Up to Date at Baseline | 43.9 | 42.0
  Up to Date at Follow Up | 66.7 | 66.8
Statistical Analysis 1: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Test type: Superiority — Test the coefficient for intervention; p = 0.8501, Regression, Logistic — Treatment Group (CCI vs PCM); p<0.05; Odds Ratio (OR) = 1.031, 95% CI 2-sided [0.753 to 1.410] — In the logistic regression model, adjustments were made for PHQ9 at baseline, improvement of depression by one level, baseline breast cancer up to date status, age, and income

4. Primary Outcome: Assessment of Cervical Cancer Screening Up to Date Status After Intervention
Description: Multivariate logistic regression model was used to assess which factors contributed to cervical cancer screening up to date status
Time Frame: Baseline - 12 months
Measure: Number; unit: Percentage of participants
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM)
Number analyzed (Participants) | 378 | 379
Percentage of participants
  Up to Date at Baseline | 42.3 | 41.7
  Up to Date at Follow Up | 61.6 | 64.6
Statistical Analysis 1: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Test type: Superiority — Test the coefficient for intervention; p = 0.4432, Regression, Logistic — Treatment Group(CCI vs PCM); p<0.05; Odds Ratio (OR) = 0.876, 95% CI 2-sided [0.625 to 1.228] — In the logistic regression model, adjustments were made for PHQ9 at baseline, improvement of depression by one level, baseline cervical cancer up to date status, age, and income

5. Primary Outcome: Comparison of Change in Patient Health Questionnaire-9 (PHQ9) Score by Intervention Arm
Description: Comparison of change in depression between the CCI and PCM arm before and after intervention. (Self-Report).
  The Patient Health Questionnaire-9 (PHQ9) is a well-validated measure of Diagnostic and Statistical Manual of Mental Disorders 4th Edition (DSM-IV) criteria for screening and diagnosing depressive episode, assessing severity, and monitoring treatment response. The PHQ9 score ranges from the minimum of 0 (no depression) to the maximum of 27 (severe depression). The detailed PHQ9 scores and corresponding level of depression severity are as follow: 0 (no depression), 1-4 (mild depression), 5-9 (medium-mild depression), 10-14 (moderate depression), 15-19 (moderately severe depression) and 20-27 (severe depression).
  The mean change in PHQ9 score is the mean of the differences between PHQ9 score at baseline and the PHQ9 score at follow up for all cases in the respective intervention arm; the greater the change in PHQ9 score, the greater the improvement in depression severity.
Time Frame: Baseline - 12 months
Population: These data are collected at baseline and 12 months. Not all participants completed all instruments at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM)
Number analyzed (Participants) | 306 | 323
units on a scale
  Mean PHQ9 Score at Baseline | 12.90 (4.22) | 12.96 (4.08)
  Mean PHQ9 Score at Follow Up | 8.24 (6.67) | 7.84 (6.24)
  Mean Change in PHQ9 Score | 4.60 (6.67) | 5.05 (6.44)
Statistical Analysis 1: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); PHQ9 Intervention Arm Difference between baseline and 12-month follow up; Test type: Superiority; p = 0.39, Two-sample t-test; p<0.05

6. Primary Outcome: Change From Baseline in The Hopkins Symptom Checklist (SCL-20) at 6 Months
Description: The SCL-20 consists of the 20 depression items on a 4-point scale from the SCL-90, and has been shown to be a valid and reliable measure of depression in diverse outpatient and community populations.
Time Frame: Baseline - 6 months
Population: This data is collected at baseline and 6 months. Not all participants completed all instruments at all time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM)
Number analyzed (Participants) | 327 | 333
Participants
  Baseline: No Depression (<0.5) | 37 | 43
  Baseline: Mild to Moderate Depression (0.5 - 1.7) | 198 | 189
  Baseline: Severe Depression (> 1.7) | 92 | 101
  6 month: number analyzed (Participants) | 292 | 300
  6 month: No Depression (<0.5) | 100 | 97
  6 month: Mild to Moderate Depression (0.5 - 1.7) | 137 | 147
  6 month: Severe Depression (> 1.7) | 55 | 56
Statistical Analysis 1: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); The Hopkins Symptom Checklist (SCL-20) at baseline; Test type: Superiority; p = 0.60, Chi-squared
Statistical Analysis 2: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); The Hopkins Symptom Checklist (SCL-20) at 6 Months; Test type: Superiority; p = 0.86, Chi-squared

7. Primary Outcome: Change From Baseline in The Hopkins Symptom Checklist (SCL-20) at 12 Months
Description: as for outcome 6
Time Frame: Baseline - 12 months
Population: This data is collected at baseline and 12 months. Not all participants completed all instruments at all time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM)
Number analyzed (Participants) | 327 | 333
Participants
  Baseline: No Depression (<0.5) | 37 | 43
  Baseline: Mild to Moderate Depression (0.5 - 1.7) | 198 | 189
  Baseline: Severe Depression (> 1.7) | 92 | 101
  12 Months: number analyzed (Participants) | 297 | 311
  12 Months: No Depression (<0.5) | 113 | 120
  12 Months: Mild to Moderate Depression (0.5 - 1.7) | 121 | 141
  12 Months: Severe Depression (> 1.7) | 63 | 50
Statistical Analysis 1: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); The Hopkins Symptom Checklist (SCL-20) at Baseline; Test type: Superiority; p = 0.60, Chi-squared
Statistical Analysis 2: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); The Hopkins Symptom Checklist (SCL-20) at 12 months; Test type: Superiority; p = 0.23, Chi-squared

8. Primary Outcome: Changes From Baseline in Number of Participants With Colorectal, Breast, and/or Cervical Cancer Screening
Description: Self-Report: We will ask participants about their participation (yes/no) in specific screening methods: Pap testing (past 3 years), mammography (past 2 years), and colorectal screening (fecal occult blood tests (FOBT)/fecal immunohistochemical tests (FIT)), past year; flexible sigmoidoscopy, the past 5 years; and colonoscopy, past 10 years).
Time Frame: Baseline - 12 months
Population: This data is collected at baseline and 12 months. Not all participants completed all instruments at all time points.
Measure: Number; unit: Percentage (%) of Participants
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM)
Number analyzed (Participants) | 378 | 379
Percentage (%) of Participants
  Colorectal Cancer Screening - Baseline | 42.9 | 44.1
  Colorectal Cancer Screening - Follow Up: number analyzed (Participants) | 316 | 333
  Colorectal Cancer Screening - Follow Up | 71.2 | 68.5
  Breast Cancer Screening - Baseline: number analyzed (Participants) | 363 | 366
  Breast Cancer Screening - Baseline | 69.2 | 72.1
  Breast Cancer Screening - Follow Up: number analyzed (Participants) | 308 | 323
  Breast Cancer Screening - Follow Up | 89.9 | 87.6
  Cervical Cancer Screening - Baseline: number analyzed (Participants) | 377 | 376
  Cervical Cancer Screening - Baseline | 83.3 | 82.2
  Cervical Cancer Screening - Follow Up: number analyzed (Participants) | 312 | 329
  Cervical Cancer Screening - Follow Up | 87.2 | 90.6
Statistical Analysis 1: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Colorectal Cancer Screening Intervention Arm Difference at 12 Months; Test type: Superiority; p = 0.4483, Chi-squared; p<0.05
Statistical Analysis 2: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Cervical Cancer Screening Intervention Arm Difference at 12 Months; Test type: Superiority; p = 0.1706, Chi-squared; p<0.05
Statistical Analysis 3: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Breast Cancer Screening Intervention Arm Difference at 12 Months; Test type: Superiority; p = 0.3568, Chi-squared; p<0.05

9. Secondary Outcome: Mental Health Care Utilization: Assessed by Patient Report
Description: Participants were asked how many times in the past six months they had seen a provider to talk about or to receive medication for feeling sad, nervous, hopeless, or blue. This question was adapted from the NCI's HINTS survey. Two categories were created using the median as a cut point. The two categories were high utilization and low utilization.
Time Frame: Baseline, 6 months and 12 months
Population: This data is collected at baseline, 6 months and 12 months for 3 different instruments. Not all participants completed all instruments at all time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM)
Number analyzed (Participants) | 378 | 379
Participants
  Mental Health Visits - Baseline: High Utilization | 162 | 165
  Mental Health Visits - Baseline: Low Utilization | 216 | 214
  Mental Health Visits - 6 Months: number analyzed (Participants) | 313 | 326
  Mental Health Visits - 6 Months: High Utilization | 116 | 136
  Mental Health Visits - 6 Months: Low Utilization | 197 | 190
  Mental Health Visits - 12 Months: number analyzed (Participants) | 316 | 333
  Mental Health Visits - 12 Months: High Utilization | 125 | 132
  Mental Health Visits - 12 Months: Low Utilization | 191 | 201
  Mental Health Prescriptions - Baseline: High Utilization | 137 | 145
  Mental Health Prescriptions - Baseline: Low Utilization | 241 | 234
  Mental Health Prescriptions - 6 Months: number analyzed (Participants) | 313 | 326
  Mental Health Prescriptions - 6 Months: High Utilization | 126 | 130
  Mental Health Prescriptions - 6 Months: Low Utilization | 187 | 196
  Mental Health Prescriptions - 12 Months: number analyzed (Participants) | 316 | 333
  Mental Health Prescriptions - 12 Months: High Utilization | 128 | 135
  Mental Health Prescriptions - 12 Months: Low Utilization | 188 | 198
Statistical Analysis 1: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Mental Health Care Utilization - Mental Health Visits at baseline; Test type: Superiority; p = 0.85, Chi-squared
Statistical Analysis 2: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Mental Health Care Utilization - Mental Health Visits at 6 months; Test type: Superiority; p = 0.23, Chi-squared
Statistical Analysis 3: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Mental Health Care Utilization - Mental Health Visits at 12 months; Test type: Superiority; p = 0.98, Chi-squared
Statistical Analysis 4: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Mental Health Care Utilization - Mental Health Prescriptions at baseline; Test type: Superiority; p = 0.57, Chi-squared
Statistical Analysis 5: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Mental Health Care Utilization - Mental Health Prescriptions at 6 months; Test type: Superiority; p = 0.92, Chi-squared
Statistical Analysis 6: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Mental Health Care Utilization - Mental Health Prescriptions at 12 months; Test type: Superiority; p = 0.99, Chi-squared

10. Secondary Outcome: Satisfaction With Decision to Participate in Screening and Mental Health Care as Assessed by Decision Scale
Description: The Satisfaction with Decision Scale is a 6-item measure that uses a five-point Likert-type scale; it is grounded in a conceptual model of an effective decision, i.e., one that is informed, consistent with the decision-maker's values, and behaviorally implemented. This scale has been tailored to healthcare decisions to receive treatment for emotional or mental health and to have cervical, breast, and colon cancer screening.The continuous summary score was converted into two categories using the median as a cut point. The two categories are high satisfaction and low satisfaction.
Time Frame: Baseline, 6 months and 12 months
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM)
Number analyzed (Participants) | 374 | 376
Participants
  Colorectal Cancer Screening - Baseline: number analyzed (Participants) | 373 | 376
  Colorectal Cancer Screening - Baseline: High Satisfaction | 161 | 180
  Colorectal Cancer Screening - Baseline: Low Satisfaction | 212 | 196
  Colorectal Cancer Screening - 6 months: number analyzed (Participants) | 295 | 301
  Colorectal Cancer Screening - 6 months: High Satisfaction | 112 | 131
  Colorectal Cancer Screening - 6 months: Low Satisfaction | 183 | 170
  Colorectal Cancer Screening - 12 months: number analyzed (Participants) | 305 | 323
  Colorectal Cancer Screening - 12 months: High Satisfaction | 135 | 148
  Colorectal Cancer Screening - 12 months: Low Satisfaction | 170 | 175
  Breast Cancer Screening - Baseline: High Satisfaction | 186 | 192
  Breast Cancer Screening - Baseline: Low Satisfaction | 188 | 184
  Breast Cancer Screening - 6 months: number analyzed (Participants) | 298 | 303
  Breast Cancer Screening - 6 months: High Satisfaction | 147 | 145
  Breast Cancer Screening - 6 months: Low Satisfaction | 151 | 158
  Breast Cancer Screening - 12 months: number analyzed (Participants) | 307 | 323
  Breast Cancer Screening - 12 months: High Satisfaction | 150 | 160
  Breast Cancer Screening - 12 months: Low Satisfaction | 157 | 163
  Cervical Cancer Screening - Baseline: number analyzed (Participants) | 295 | 294
  Cervical Cancer Screening - Baseline: High Satisfaction | 147 | 152
  Cervical Cancer Screening - Baseline: Low Satisfaction | 148 | 142
  Cervical Cancer Screening - 6 months: number analyzed (Participants) | 221 | 231
  Cervical Cancer Screening - 6 months: High Satisfaction | 99 | 101
  Cervical Cancer Screening - 6 months: Low Satisfaction | 122 | 130
  Cervical Cancer Screening - 12 Months: number analyzed (Participants) | 226 | 251
  Cervical Cancer Screening - 12 Months: High Satisfaction | 107 | 120
  Cervical Cancer Screening - 12 Months: Low Satisfaction | 119 | 131
  Mental Health Care - 12 Months: number analyzed (Participants) | 304 | 319
  Mental Health Care - 12 Months: High Satisfaction | 129 | 128
  Mental Health Care - 12 Months: Low Satisfaction | 175 | 191
Statistical Analysis 1: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Satisfaction with decision to participate in colorectal cancer screening at baseline; Test type: Superiority; p = 0.20, Chi-squared
Statistical Analysis 2: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Satisfaction with decision to participate in colorectal cancer screening at 6 months; Test type: Superiority; p = 0.17, Chi-squared
Statistical Analysis 3: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Satisfaction with decision to participate in colorectal cancer screening at 12 months; Test type: Superiority; p = 0.69, Chi-squared
Statistical Analysis 4: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Satisfaction with decision to participate in breast cancer screening at baseline; Test type: Superiority; p = 0.72, Chi-squared
Statistical Analysis 5: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Satisfaction with decision to participate in breast cancer screening at 6 months; Test type: Superiority; p = 0.72, Chi-squared
Statistical Analysis 6: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Satisfaction with decision to participate in breast cancer screening at 12 months; Test type: Superiority; p = 0.87, Chi-squared
Statistical Analysis 7: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Satisfaction with decision to participate in cervical cancer screening at baseline; Test type: Superiority; p = 0.65, Chi-squared
Statistical Analysis 8: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Satisfaction with decision to participate in cervical cancer screening at 6 months; Test type: Superiority; p = 0.82, Chi-squared
Statistical Analysis 9: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Satisfaction with decision to participate in cervical cancer screening at 12 months; Test type: Superiority; p = 0.92, Chi-squared
Statistical Analysis 10: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Satisfaction with decision to participate in Mental Health Care at 12 months; Test type: Superiority; p = 0.56, Chi-squared

11. Secondary Outcome: Physician Recommendation of Screening/Mental Health Care
Description: This questionnaire, adopted from National Cancer Institute's (NCI) Health Information National Trends Survey (HINTS), assesses whether patients report that their primary care physician 1) has recommended cervical, breast, and colon cancer screening and 2) has recommended that the patient make an appointment with a mental health provider and/or take psychotropic medication. Two categories were created according to whether the patient received a physician recommendation (yes/no). The category of "Recommendation" for when they received a recommendation and a category of "No Recommendation" if they did not receive a recommendation
Time Frame: Baseline, 6 months and 12 months
Population: Data are collected at baseline, 6 months and 12 months. Not all participants completed the assessment at all time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM)
Number analyzed (Participants) | 378 | 379
Participants
  Colorectal Cancer Screening - Baseline: number analyzed (Participants) | 378 | 378
  Colorectal Cancer Screening - Baseline: Recommendation | 298 | 282
  Colorectal Cancer Screening - Baseline: No Recommendation | 80 | 96
  Colorectal Cancer Screening - 6 Months: number analyzed (Participants) | 304 | 314
  Colorectal Cancer Screening - 6 Months: Recommendation | 281 | 284
  Colorectal Cancer Screening - 6 Months: No Recommendation | 23 | 30
  Colorectal Cancer Screening - 12 Months: number analyzed (Participants) | 312 | 328
  Colorectal Cancer Screening - 12 Months: Recommendation | 281 | 308
  Colorectal Cancer Screening - 12 Months: No Recommendation | 31 | 20
  Breast Cancer Screening - Baseline: number analyzed (Participants) | 377 | 376
  Breast Cancer Screening - Baseline: Recommendation | 340 | 339
  Breast Cancer Screening - Baseline: No Recommendation | 37 | 37
  Breast Cancer Screening - 6 Months: number analyzed (Participants) | 304 | 314
  Breast Cancer Screening - 6 Months: Recommendation | 299 | 303
  Breast Cancer Screening - 6 Months: No Recommendation | 5 | 11
  Breast Cancer Screening - 12 Months: number analyzed (Participants) | 312 | 329
  Breast Cancer Screening - 12 Months: Recommendation | 302 | 321
  Breast Cancer Screening - 12 Months: No Recommendation | 10 | 8
  Cervical Cancer Screening - Baseline: number analyzed (Participants) | 378 | 376
  Cervical Cancer Screening - Baseline: Recommendation | 309 | 297
  Cervical Cancer Screening - Baseline: No Recommendation | 69 | 79
  Cervical Cancer Screening - 6 Months: number analyzed (Participants) | 304 | 314
  Cervical Cancer Screening - 6 Months: Recommendation | 281 | 283
  Cervical Cancer Screening - 6 Months: No Recommendation | 23 | 31
  Cervical Cancer Screening - 12 Months: number analyzed (Participants) | 312 | 327
  Cervical Cancer Screening - 12 Months: Recommendation | 279 | 299
  Cervical Cancer Screening - 12 Months: No Recommendation | 33 | 28
  Mental Health Care - Baseline: number analyzed (Participants) | 378 | 374
  Mental Health Care - Baseline: Recommendation | 206 | 206
  Mental Health Care - Baseline: No Recommendation | 172 | 168
  Mental Health Care - 6 Months: number analyzed (Participants) | 304 | 313
  Mental Health Care - 6 Months: Recommendation | 183 | 191
  Mental Health Care - 6 Months: No Recommendation | 121 | 122
  Mental Health Care - 12 Months: number analyzed (Participants) | 312 | 328
  Mental Health Care - 12 Months: Recommendation | 182 | 203
  Mental Health Care - 12 Months: No Recommendation | 130 | 125
Statistical Analysis 1: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Physician Recommendation of Colorectal Cancer Screening at baseline; Test type: Superiority; p = 0.17, Chi-squared
Statistical Analysis 2: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Physician Recommendation of Colorectal Cancer Screening at 6 months; Test type: Superiority; p = 0.38, Chi-squared
Statistical Analysis 3: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Physician Recommendation of Colorectal Cancer Screening at 12 months; Test type: Superiority; p = 0.07, Chi-squared
Statistical Analysis 4: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Physician Recommendation of Breast Cancer Screening at baseline; Test type: Superiority; p = 0.99, Chi-squared
Statistical Analysis 5: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Physician Recommendation of Breast Cancer Screening at 6 months; Test type: Superiority; p = 0.15, Chi-squared
Statistical Analysis 6: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Physician Recommendation of Breast Cancer Screening at 12 months; Test type: Superiority; p = 0.55, Chi-squared
Statistical Analysis 7: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Physician Recommendation of Cervical Cancer Screening at baseline; Test type: Superiority; p = 0.34, Chi-squared
Statistical Analysis 8: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Physician Recommendation of Cervical Cancer Screening at 6 months; Test type: Superiority; p = 0.31, Chi-squared
Statistical Analysis 9: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Physician Recommendation of Cervical Cancer Screening at 12 months; Test type: Superiority; p = 0.39, Chi-squared
Statistical Analysis 10: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Physician Recommendation of Mental Health Care at baseline; Test type: Superiority; p = 0.87, Chi-squared
Statistical Analysis 11: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Physician Recommendation of Mental Health Care at 6 months; Test type: Superiority; p = 0.83, Chi-squared
Statistical Analysis 12: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Physician Recommendation of Mental Health Care at 12 months; Test type: Superiority; p = 0.36, Chi-squared

12. Secondary Outcome: Generalized Anxiety Disorder
Description: This Generalized Anxiety Disorder scale is based on diagnostic criteria in the Diagnostic and Statistical Manual of Mental Disorders 4th Edition (DSM-IV) and measures probable anxiety disorder and severity of anxiety symptoms. Patients are asked to rate how often they have been bothered by 7 problems in the last 2 weeks on a 4-point scale. Standard cut points were used for the Generalized Anxiety Disorder measure. Minimal anxiety is (0-4). Mild Anxiety would be count as (5-9). Moderate Anxiety (10-14) and severe anxiety would be (15-21).
Time Frame: Baseline, 6 months and 12 months
Population: This data is collected at baseline, 6 months and 12 months. Not all participants completed the assessment at all time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM)
Number analyzed (Participants) | 372 | 372
Participants
  Baseline: Minimal Anxiety (0-4) | 79 | 79
  Baseline: Mild Anxiety (5-9) | 114 | 108
  Baseline: Moderate Anxiety (10-14) | 89 | 95
  Baseline: Severe Anxiety (15-21) | 90 | 90
  6 months: number analyzed (Participants) | 300 | 301
  6 months: Minimal Anxiety (0-4) | 133 | 127
  6 months: Mild Anxiety (5-9) | 69 | 82
  6 months: Moderate Anxiety (10-14) | 61 | 42
  6 months: Severe Anxiety (15-21) | 37 | 50
  12 months: number analyzed (Participants) | 308 | 322
  12 months: Minimal Anxiety (0-4) | 124 | 145
  12 months: Mild Anxiety (5-9) | 82 | 77
  12 months: Moderate Anxiety (10-14) | 46 | 56
  12 months: Severe Anxiety (15-21) | 56 | 44
Statistical Analysis 1: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Generalized Anxiety Disorder scale at baseline. Coding of the measure was based on Spitzer, R.L., Kroenke, K., Williams, J.B., & Lowe, B. (2006); Test type: Superiority; p = 0.95, Chi-squared
Statistical Analysis 2: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Generalized Anxiety Disorder scale score at 6 months. Coding of the measure was based on Spitzer, R.L., Kroenke, K., Williams, J.B., & Lowe, B. (2006); Test type: Superiority; p = 0.08, Chi-squared
Statistical Analysis 3: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Generalized Anxiety Disorder scale score at 12 months. Coding of the measure was based on Spitzer, R.L., Kroenke, K., Williams, J.B., & Lowe, B. (2006); Test type: Superiority; p = 0.27, Chi-squared

13. Secondary Outcome: Medical Outcomes Study Health Survey-Short Form
Description: The quality of life was measured with the Medical Outcomes Study (MOS) Short Form Health Survey (SF-12) is a general measure of health status that assess the patient's perceived health status and whether health problems interfere with normal functioning. The SF-12 has demonstrated validity and test-retest reliability in the general population and in patients with chronic health conditions, and has been tested in five languages, including Spanish. It has been used extensively as a quality of life measure in collaborative care studies, including with low-income minority populations. It has also been used frequently in screening studies, for cancer and other conditions. The SF-12 has been validated as an indicator of effects of depression on quality of life in ethnically diverse patients.
  The continuous summary score was converted into 4 categories using quartiles as cutoff points. The four categories are Best Health, Good health, Fair Health and Worst Health.
Time Frame: Baseline, 6 months and 12 months
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM)
Number analyzed (Participants) | 370 | 359
Participants
  Baseline: Best Health | 96 | 88
  Baseline: Good Health | 86 | 95
  Baseline: Fair Health | 92 | 96
  Baseline: Worst Health | 96 | 80
  6 months: number analyzed (Participants) | 293 | 302
  6 months: Best Health | 70 | 74
  6 months: Good Health | 77 | 82
  6 months: Fair Health | 65 | 75
  6 months: Worst Health | 81 | 71
  12 months: number analyzed (Participants) | 307 | 319
  12 months: Best Health | 73 | 83
  12 months: Good Health | 79 | 77
  12 months: Fair Health | 72 | 83
  12 months: Worst Health | 83 | 76
Statistical Analysis 1: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Medical Outcomes Study Health Survey at baseline. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.54, Chi-squared
Statistical Analysis 2: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Medical Outcomes Study Health Survey at 6 months. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.68, Chi-squared
Statistical Analysis 3: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Medical Outcomes Study Health Survey at 12 months. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.68, Chi-squared

14. Secondary Outcome: Breast, Cervical and Colorectal Cancer Screening Attitudes
Description: This measure was adapted from the National Cancer Institute's HINTS questions for colorectal cancer.
  The continuous summary score was converted into 4 categories using quartiles as cut points. The categories for screening attitudes were as follows: positive attitudes, moderate attitudes, fair attitudes and negative attitudes.
Time Frame: Baseline, 6 months and 12 months
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM)
Number analyzed (Participants) | 377 | 377
Participants
  Colorectal Cancer Screening - Baseline: number analyzed (Participants) | 372 | 373
  Colorectal Cancer Screening - Baseline: Positive Attitudes | 71 | 71
  Colorectal Cancer Screening - Baseline: Moderate Attitudes | 45 | 55
  Colorectal Cancer Screening - Baseline: Fair Attitudes | 161 | 152
  Colorectal Cancer Screening - Baseline: Negative Attitudes | 95 | 95
  Colorectal Cancer Screening - 6 months: number analyzed (Participants) | 300 | 300
  Colorectal Cancer Screening - 6 months: Positive Attitudes | 65 | 64
  Colorectal Cancer Screening - 6 months: Moderate Attitudes | 46 | 39
  Colorectal Cancer Screening - 6 months: Fair Attitudes | 83 | 86
  Colorectal Cancer Screening - 6 months: Negative Attitudes | 106 | 111
  Colorectal Cancer Screening - 12 months: number analyzed (Participants) | 308 | 323
  Colorectal Cancer Screening - 12 months: Positive Attitudes | 131 | 134
  Colorectal Cancer Screening - 12 months: Moderate Attitudes | 0 | 0
  Colorectal Cancer Screening - 12 months: Fair Attitudes | 0 | 0
  Colorectal Cancer Screening - 12 months: Negative Attitudes | 177 | 189
  Breast Cancer Screening - Baseline: Positive Attitudes | 71 | 79
  Breast Cancer Screening - Baseline: Moderate Attitudes | 62 | 61
  Breast Cancer Screening - Baseline: Fair Attitudes | 136 | 132
  Breast Cancer Screening - Baseline: Negative Attitudes | 108 | 105
  Breast Cancer Screening - 6 months: number analyzed (Participants) | 300 | 306
  Breast Cancer Screening - 6 months: Positive Attitudes | 126 | 124
  Breast Cancer Screening - 6 months: Moderate Attitudes | 0 | 0
  Breast Cancer Screening - 6 months: Fair Attitudes | 0 | 0
  Breast Cancer Screening - 6 months: Negative Attitudes | 174 | 182
  Breast Cancer Screening - 12 months: number analyzed (Participants) | 308 | 325
  Breast Cancer Screening - 12 months: Positive Attitudes | 131 | 142
  Breast Cancer Screening - 12 months: Moderate Attitudes | 0 | 0
  Breast Cancer Screening - 12 months: Fair Attitudes | 0 | 0
  Breast Cancer Screening - 12 months: Negative Attitudes | 177 | 183
  Cervical Cancer Screening - Baseline: number analyzed (Participants) | 300 | 295
  Cervical Cancer Screening - Baseline: Positive Attitudes | 60 | 64
  Cervical Cancer Screening - Baseline: Moderate Attitudes | 51 | 58
  Cervical Cancer Screening - Baseline: Fair Attitudes | 107 | 92
  Cervical Cancer Screening - Baseline: Negative Attitudes | 82 | 81
  Cervical Cancer Screening - 6 months: number analyzed (Participants) | 223 | 230
  Cervical Cancer Screening - 6 months: Positive Attitudes | 99 | 85
  Cervical Cancer Screening - 6 months: Moderate Attitudes | 0 | 0
  Cervical Cancer Screening - 6 months: Fair Attitudes | 0 | 0
  Cervical Cancer Screening - 6 months: Negative Attitudes | 124 | 145
  Cervical Cancer Screening - 12 months: number analyzed (Participants) | 227 | 250
  Cervical Cancer Screening - 12 months: Positive Attitudes | 98 | 108
  Cervical Cancer Screening - 12 months: Moderate Attitudes | 0 | 0
  Cervical Cancer Screening - 12 months: Fair Attitudes | 0 | 0
  Cervical Cancer Screening - 12 months: Negative Attitudes | 129 | 142
Statistical Analysis 1: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Colorectal Cancer Screening attitudes at baseline. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.74, Chi-squared
Statistical Analysis 2: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Colorectal Cancer Screening attitudes at 6 months. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.86, Chi-squared
Statistical Analysis 3: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Colorectal Cancer Screening attitudes at 12 months. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.79, Chi-squared
Statistical Analysis 4: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Breast Cancer Screening attitudes at baseline. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.91, Chi-squared
Statistical Analysis 5: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Breast Cancer Screening attitudes at 6 months. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.71, Chi-squared
Statistical Analysis 6: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Breast Cancer Screening attitudes at 12 months. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.77, Chi-squared
Statistical Analysis 7: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Cervical Cancer Screening attitudes at baseline. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.64, Chi-squared
Statistical Analysis 8: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Cervical Cancer Screening attitudes at 6 months. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.11, Chi-squared
Statistical Analysis 9: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Cervical Cancer Screening attitudes at 12 months. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 1.00, Chi-squared

15. Secondary Outcome: Satisfaction With Decision Scale- Cancer Screening (Data Reported in Outcome Measure #10)
Description: The Satisfaction with Decision Scale is a 6-item measure that uses a five-point Likert-type scale; it is grounded in a conceptual model of an effective decision, i.e., one that is informed, consistent with the decision-maker's values, and behaviorally implemented. This scale has been tailored to healthcare decisions to have cervical, breast, and colon cancer screening.The satisfaction with decision scale of cancer screening and its continuous summary score was converted into two categories (high satisfaction and low satisfaction) using the median as the cutoff point.
Time Frame: Baseline, 6 months and 12 months
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM)
Number analyzed (Participants) | 373 | 376
Participants
  Colorectal Cancer Screening - Baseline: High Satisfaction | 161 | 180
  Colorectal Cancer Screening - Baseline: Low Satisfaction | 212 | 196
  Colorectal Cancer Screening - 6 months: number analyzed (Participants) | 295 | 301
  Colorectal Cancer Screening - 6 months: High Satisfaction | 112 | 131
  Colorectal Cancer Screening - 6 months: Low Satisfaction | 183 | 170
  Colorectal Cancer Screening - 12 Months: number analyzed (Participants) | 305 | 323
  Colorectal Cancer Screening - 12 Months: High Satisfaction | 135 | 148
  Colorectal Cancer Screening - 12 Months: Low Satisfaction | 170 | 175

16. Secondary Outcome: Satisfaction With Decision Scale- Mental Health (Data Reported in Secondary Outcome Measure #10)
Description: The Satisfaction with Decision Scale is a 6-item measure that uses a five-point Likert-type scale; it is grounded in a conceptual model of an effective decision, i.e., one that is informed, consistent with the decision-maker's values, and behaviorally implemented. This scale has been tailored to healthcare decisions to have mental health care.The satisfaction with decision scale of mental health and its continuous summary score was converted into two categories (high satisfaction and low satisfaction) using the median as the cutoff point.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM)
Number analyzed (Participants) | 304 | 319
Participants
  High Satisfaction | 129 | 128
  Low Satisfaction | 175 | 191
Statistical Analysis 1: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Satisfaction with decision to participate in Mental Health Care at 12 months. Recoding of the continuous measure was based on quartiles; Test type: Superiority; p = 0.56, Chi-squared

17. Secondary Outcome: Devaluation-Discrimination Scale
Description: This measure was adapted from the Link's Devaluation-Discrimination Scale.The continuous summary score was converted into 4 categories using quartiles as cut points. The 4 categories were as follows: Low stigma, minimal stigma, moderate stigma and high stigma.
Time Frame: Baseline and 12 months
Population: This data is collected at baseline and 12 months. Not all participants completed this instrument at all time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM)
Number analyzed (Participants) | 192 | 193
Participants
  Baseline: Low Stigma | 68 | 50
  Baseline: Minimal Stigma | 42 | 45
  Baseline: Moderate Stigma | 46 | 49
  Baseline: High Stigma | 36 | 49
  12 months: number analyzed (Participants) | 160 | 163
  12 months: Low Stigma | 50 | 55
  12 months: Minimal Stigma | 36 | 48
  12 months: Moderate Stigma | 30 | 26
  12 months: High Stigma | 44 | 34
Statistical Analysis 1: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Devaluation-Discrimination Scale Score at baseline. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.18, Chi-squared
Statistical Analysis 2: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Devaluation-Discrimination Scale score at 12 months. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.32, Chi-squared

18. Secondary Outcome: Ambulatory Care Experiences as Assessed by Ambulatory Care Experiences Survey
Description: The Ambulatory Care Experiences Survey produces 11 summary measures covering 2 broad dimensions of patients' experiences: quality of physician-patient interactions and organizational features of care.
  The continuous summary score was converted into 4 categories (High, Moderate, Fair and Low) using quartiles as cut-points.
Time Frame: Baseline, 6 months and 12 months
Population: This data is collected at baseline, 6 months and 12 months. Not all participants completed this instrument at all time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM)
Number analyzed (Participants) | 378 | 379
Participants
  Shared Decision Making - Baseline: High | 114 | 123
  Shared Decision Making - Baseline: Moderate | 0 | 0
  Shared Decision Making - Baseline: Fair | 0 | 0
  Shared Decision Making - Baseline: Low | 264 | 256
  Shared Decision Making - 6 Months: number analyzed (Participants) | 313 | 326
  Shared Decision Making - 6 Months: High | 81 | 77
  Shared Decision Making - 6 Months: Moderate | 0 | 0
  Shared Decision Making - 6 Months: Fair | 0 | 0
  Shared Decision Making - 6 Months: Low | 232 | 249
  Shared Decision Making - 12 Months: number analyzed (Participants) | 316 | 333
  Shared Decision Making - 12 Months: High | 77 | 108
  Shared Decision Making - 12 Months: Moderate | 0 | 0
  Shared Decision Making - 12 Months: Fair | 0 | 0
  Shared Decision Making - 12 Months: Low | 239 | 225
  Access - Baseline: High | 24 | 23
  Access - Baseline: Moderate | 25 | 22
  Access - Baseline: Fair | 23 | 27
  Access - Baseline: Low | 306 | 307
  Access - 6 Months: number analyzed (Participants) | 313 | 326
  Access - 6 Months: High | 26 | 30
  Access - 6 Months: Moderate | 0 | 0
  Access - 6 Months: Fair | 0 | 0
  Access - 6 Months: Low | 287 | 296
  Access - 12 Months: number analyzed (Participants) | 316 | 333
  Access - 12 Months: High | 28 | 26
  Access - 12 Months: Moderate | 0 | 0
  Access - 12 Months: Fair | 0 | 0
  Access - 12 Months: Low | 288 | 307
  Care Coordination - Baseline: High | 67 | 61
  Care Coordination - Baseline: Moderate | 0 | 0
  Care Coordination - Baseline: Fair | 0 | 0
  Care Coordination - Baseline: Low | 311 | 318
  Care Coordination - 6 Months: number analyzed (Participants) | 313 | 326
  Care Coordination - 6 Months: High | 30 | 19
  Care Coordination - 6 Months: Moderate | 22 | 22
  Care Coordination - 6 Months: Fair | 23 | 27
  Care Coordination - 6 Months: Low | 238 | 258
  Care Coordination - 12 Months: number analyzed (Participants) | 316 | 333
  Care Coordination - 12 Months: High | 18 | 26
  Care Coordination - 12 Months: Moderate | 9 | 4
  Care Coordination - 12 Months: Fair | 39 | 31
  Care Coordination - 12 Months: Low | 250 | 272
  Quality - Baseline: High | 142 | 152
  Quality - Baseline: Moderate | 0 | 0
  Quality - Baseline: Fair | 0 | 0
  Quality - Baseline: Low | 236 | 227
  Quality - 6 Months: number analyzed (Participants) | 313 | 326
  Quality - 6 Months: High | 121 | 115
  Quality - 6 Months: Moderate | 0 | 0
  Quality - 6 Months: Fair | 0 | 0
  Quality - 6 Months: Low | 192 | 211
  Quality - 12 Months: number analyzed (Participants) | 316 | 333
  Quality - 12 Months: High | 116 | 122
  Quality - 12 Months: Moderate | 0 | 0
  Quality - 12 Months: Fair | 0 | 0
  Quality - 12 Months: Low | 200 | 211
Statistical Analysis 1: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Ambulatory Care Experiences - Shared Decision Making at baseline. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.50, Chi-squared
Statistical Analysis 2: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Ambulatory Care Experiences - Shared Decision Making at six months. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.51, Chi-squared
Statistical Analysis 3: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Ambulatory Care Experiences - Shared Decision Making at twelve months. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.02, Chi-squared
Statistical Analysis 4: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Ambulatory Care Experiences - Access at baseline. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.91, Chi-squared
Statistical Analysis 5: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Ambulatory Care Experiences - Access at six months. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.69, Chi-squared
Statistical Analysis 6: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Ambulatory Care Experiences - Access at twelve months. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.63, Chi-squared
Statistical Analysis 7: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Ambulatory Care Experiences - Care Coordination at baseline. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.55, Chi-squared
Statistical Analysis 8: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Ambulatory Care Experiences - Care Coordination at six months. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.34, Chi-squared
Statistical Analysis 9: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Ambulatory Care Experiences - Care Coordination at twelve months. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.19, Chi-squared
Statistical Analysis 10: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Ambulatory Care Experiences - Quality at baseline. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.47, Chi-squared
Statistical Analysis 11: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Ambulatory Care Experiences - Quality at six months. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.38, Chi-squared
Statistical Analysis 12: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Ambulatory Care Experiences - Quality at twelve months. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.98, Chi-squared

19. Secondary Outcome: Medication Adherence
Description: In this questionnaire, respondents were asked if they had been prescribed medication for depression and about difficulties taking medication(s) regularly.
  Standard cut points was used for medical adherence. High adherence- around an 8. Medium adherence - 6-7.99. Low adherence would be anything less than 6.
Time Frame: Baseline, 6 months and 12 months
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM)
Number analyzed (Participants) | 125 | 131
Participants
  Baseline: High Adherence (8) | 20 | 25
  Baseline: Medium Adherence (6-7.99) | 30 | 32
  Baseline: Low Adherence (<6) | 75 | 74
  6 months: number analyzed (Participants) | 115 | 114
  6 months: High Adherence (8) | 20 | 23
  6 months: Medium Adherence (6-7.99) | 35 | 23
  6 months: Low Adherence (<6) | 60 | 68
  12 months: number analyzed (Participants) | 115 | 119
  12 months: High Adherence (8) | 22 | 27
  12 months: Medium Adherence (6-7.99) | 33 | 31
  12 months: Low Adherence (<6) | 60 | 61
Statistical Analysis 1: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Medication Adherence at baseline. Coding of the measure was based on Morisky et al. (2008); Test type: Superiority; p = 0.78, Chi-squared
Statistical Analysis 2: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Medication Adherence at 6 months. Coding of the measure was based on Morisky et al. (2008); Test type: Superiority; p = 0.20, Chi-squared
Statistical Analysis 3: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Medication Adherence at 12 Months. Coding of the measure was based on Morisky et al. (2008); Test type: Superiority; p = 0.77, Chi-squared

20. Secondary Outcome: Self-efficacy and Behavior Towards Cancer Screening/Mental Health Utilization
Description: This 5-item scale measures a sense of perceived self-efficacy associated with accessing and paying for the three different types of cancer screening and utilization of needed mental health services.
  The continuous study score was converted into 4 categories using quartiles as cut points. The 4 categories are high self-efficacy, moderate self- efficacy, minimal self-efficacy and low self-efficacy.
Time Frame: Baseline, 6 months and 12 months
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM)
Number analyzed (Participants) | 373 | 373
Participants
  Baseline: High Self-Efficacy | 98 | 87
  Baseline: Moderate Self-Efficacy | 87 | 98
  Baseline: Minimal Self-Efficacy | 90 | 87
  Baseline: Low Self-Efficacy | 98 | 101
  6 months: number analyzed (Participants) | 298 | 304
  6 months: High Self-Efficacy | 70 | 74
  6 months: Moderate Self-Efficacy | 68 | 76
  6 months: Minimal Self-Efficacy | 77 | 74
  6 months: Low Self-Efficacy | 83 | 80
  12 months: number analyzed (Participants) | 306 | 324
  12 months: High Self-Efficacy | 71 | 79
  12 months: Moderate Self-Efficacy | 81 | 81
  12 months: Minimal Self-Efficacy | 77 | 79
  12 months: Low Self-Efficacy | 77 | 85
Statistical Analysis 1: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Self-efficacy at baseline.Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.70, Chi-squared
Statistical Analysis 2: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Self-efficacy at 6 months. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.89, Chi-squared
Statistical Analysis 3: Comparison: Collaborative Care Intervention (CCI) vs Prevention Care Management (PCM); Self-efficacy at 12 months. Continuous summary score was converted into 4 categories using quartiles as cut-points; Test type: Superiority; p = 0.95, Chi-squared

ADVERSE EVENTS:
Time Frame: The adverse event data were collected over the 12 month period in which participants were followed.
Arm/Group | Collaborative Care Intervention (CCI) | Prevention Care Management (PCM) Intervention
All-Cause Mortality (participants affected / at risk) | 5/378 | 1/379
Serious Adverse Events (participants affected / at risk) | 1/378 | 0/379
Other Adverse Events (participants affected / at risk) | 4/378 | 4/379
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Collaborative Care Intervention (CCI) (N=378) | Prevention Care Management (PCM) Intervention (N=379)
Stroke (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Collaborative Care Intervention (CCI) (N=378) | Prevention Care Management (PCM) Intervention (N=379)
Suicidal Ideation (Psychiatric disorders) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT02273206/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT02273206/SAP_001.pdf